CLINICAL TRIAL: NCT02625792
Title: Role of Hemostatic Powder (Endo-clotTM) in Prevention of Bleeding Within High Risk Patients After ESD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4-2015-0925
Record Dates: First submitted 2015-12-06; First posted 2015-12-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Iatrogenic Ulcer After ESD
Keywords: Post ESD ulcer; Bleeding; Prophylaxis
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endo-Clot(TM) (Experimental): The intervention group
  Interventions: Drug: Endo-Clot(TM)

INTERVENTIONS:
Drug: Endo-Clot(TM) — After patients treated with ESD, Hemostatic power was applied on the post-resection surface by Endo-Clot™ system. And treated with proton pump inhibitor as usual.

SUMMARY:
SD has become a standard treatment of gastric neoplasm confined to mucosa(epithelium). But after procedure, formation of iatrogenic gastric ulcer is inevitable. And Post ESD ulcer bleeding rate reported about 5% ~ 10% of all cases. Antiplatelet or anti-coagulation treatment might be associated higher incidence of rebleeding after ESD and iatrogenic ulcer bigger than 40mm in size is also associated.

Though several previous study have failed to show efficacy of 2nd look EGD, but those reports pointed out that visible vessels with current bleeding or highly suspect of recent bleeding (Forrest type IA~IIB) was observed about 10~20% of patients. Such patients are at high risk of bleeding.

So, Investigators hypothesize that appliance of Endo-Clot(TM) at post ESD ulcer have a significant role of protection from gastric acidic juice and help mucosa heal earlier. Thus visible vessels with risk of bleeding is going to be rarely observed at 2nd look EGD. And finally this protective effect might have an effect for prophylaxis of post ESD ulcer bleeding.

ELIGIBILITY:
Inclusion Criteria:

A. Older than 19 years old and younger than 80 years old B. Pathologically confirmed gastric adenoma and/or early gastric cancer C. Iatrogenic gastric ulcer after ESD(Endoscopic submucosal dissection) more than 40mm (at prediction) D. Patients who is taking medication such at aspirin and/or coumadin (and other anti-coagulation medication) E. ECOG performance status 0 or 1 F. Adequate renal function (serum creatinine < 1.5 mg/dL or calculated creatinine clearance ≥ 60 ml/min) G. Adequate liver function (total bilirubin < 1.5 X the upper limits of normal (ULN), AST and ALT <3 X UNL, and alkaline phosphatases < 3 X ULN or < 5 x ULN in case of liver involvement) H. Adequate BM function (WBC ≥ 3,500/µl, absolute neutrophil cell count ≥ 1,500 /µl, platelet count ≥ 100,000/µl) I. Subjects who given written informed consent after being given a full description of the study

Exclusion Criteria:

A. Previously treated by radical gastrectomy B. Adverse effect on this medication C. Pregnant or on breast feeding D. Patients who are unwilling or unable to provide informed consent, such as those with psychiatric problem, drug abuse or alcoholism

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
the bleeding rate until 4 weeks after ESD | POD ~ 4 weeks
  Post-ESD bleeding was defined by clinical symptoms or laboratory findings. Clinical symptoms such as melena or hematemesis were defined as bleeding signs.

SECONDARY OUTCOMES:
Forrest classification of the post-resection ulcer at 48 hours after ESD | POD 2
  On POD 2, patients underwent scheduled second-look endoscopy 48 hours after ESD. The artificial ulcer induced by ESD was evaluated and classified according to the Forrest classification.
the bleeding rates according to timing and subgroup | POD 0 ~ 4 weeks
  the bleeding rate until 4 weeks after ESD: Post-ESD bleeding was defined by clinical symptoms or laboratory findings. Clinical symptoms such as melena or hematemesis were defined as bleeding signs. (Acute bleeding: within 48 hours after ESD & Delayed bleeding: beyond 48 hours after ESD)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei university of medical center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be not shared and used only for this study

REFERENCES:
- [Derived] Hahn KY, Park JC, Lee YK, Shin SK, Lee SK, Lee YC. Efficacy of hemostatic powder in preventing bleeding after gastric endoscopic submucosal dissection in high-risk patients. J Gastroenterol Hepatol. 2018 Mar;33(3):656-663. doi: 10.1111/jgh.13990. PMID 28910851